CLINICAL TRIAL: NCT00530283
Title: The Clinical Utility of PET-CT in the Management of Squamous Cell Carcinoma of the Neck Nodes With Unknown Primary Malignancy
Brief Title: PET-CT for Squamous Cell Carcinoma (SCC) of the Neck Nodes Unknown Primary Malignancy
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Calgary Health Region (Other); University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: 20682
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2011-08

CONDITIONS: Squamous Cell Cancer
Keywords: Squamous; Unknown Primary; Patients with Squamous cell cancer neck nodes
MeSH Terms: conditions — Neoplasms, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients with Squamous cell cancer of neck nodes, unknown primary
  Interventions: Other: PET-CT

INTERVENTIONS:
Other: PET-CT

SUMMARY:
Patients with squamous cell cancer of neck nodes but unknown primary will have a PET-CT scan prior to biopsies. The utility of PET-CT will be determined in this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* squamous cell cancer of neck nodes with unknown primary site

Exclusion Criteria:

* unable to tolerate PET-CT
* unable to undergo examination under anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold Lau, M.D., Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada